CLINICAL TRIAL: NCT00124878
Title: Trial of Male Circumcision: HIV, STD and Behavioral Effects in Men, Women and the Community
Brief Title: Trial of Male Circumcision: HIV, Sexually Transmitted Disease (STD) and Behavioral Effects in Men, Women and the Community
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wawer, Maria J., M.D. (Individual)
Collaborators: MRC/UVRI and LSHTM Uganda Research Unit (Other); Rakai Health Sciences Program (Other); Johns Hopkins Bloomberg School of Public Health (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22006
Record Dates: First submitted 2005-07-25; First posted 2005-07-28 (Estimated); Last update posted 2007-08-10 (Estimated); Status verified 2005-07

CONDITIONS: HIV Infections; Sexually Transmitted Diseases; Papillomavirus Infections; Genital Herpes; Gonorrhea; Chlamydia Infections; Syphilis; Bacterial Vaginosis
Keywords: HIV; STDs; Male circumcision; HIV+ males; HIV-negative males; Female partners; STDs such as the following:; HPV; HSV-2; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Papillomavirus Infections; Herpes Genitalis; Gonorrhea; Chlamydia Infections; Syphilis; Vaginosis, Bacterial | interventions — Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 Male circumcision (Active Comparator): Men receive circumcision after randomization; procedure is generally provided within two weeks. A man randomized to the intervention arm who then declines circumcision for 6 or more months is considered a cross over.
  Interventions: Procedure: Male circumcision
- Arm 2 (No Intervention): Men wait for two years of follow up before being offered male circumcision
  Interventions: Procedure: Male circumcision

INTERVENTIONS:
Procedure: Male circumcision — Sleeve circumcision

SUMMARY:
This randomized controlled trial conducted in Rakai District, Uganda, has enrolled 997 HIV positive men and 500 men who declined to learn HIV results (regardless of HIV status). The hypotheses are that male circumcision will be acceptable to and safe in both groups and will reduce the rates of STD acquisition in both groups and of HIV acquisition in HIV-negative men.

Enrollment was ended on Dec 12, 2006, following an interim Data Monitoring and Safety Board (DSMB) review of a closed report. At that time the DSMB determined that futility with respect to the female HIV outcome. There was an non-significantly higher rate of HIV acquisition in women partners of HIV+ men in couples who had resumed sex prior to certified post-surgical wound healing. The data indicated significant reductions (~50%) in GUD symptoms among circumcised HIV+ men. The DSMB recommended: 1) that men and women should continue to be followed in complete two year follow up on all, 2) that circumcision for remaining HIV+ intervention arm men and for control arm men who had completed their 2 year follow should continue, contingent on a) revision of the study protocol to add additional post-surgical visits to assess wound healing, b) protocol revision to further strengthen education for both male and female partners on the need to postpone sex until certified wound healing, and c) approval of the revised protocol by the IRBs in both the US and Uganda. 3) An additional follow up visit for women be instituted at 18 months after enrollment. Protocol revision and IRB approvals have been finalized in June, 2007.

The study has also enrolled and is following 3,700 women sexual partners of men enrolled in this study and in a complementary National Institutes of Health (NIH) funded study (U1 AI51171 which is separately registered). The hypotheses are that male circumcision will be acceptable to and safe in women partners, and will reduce the women's acquisition of HIV and STDs such as herpes simplex virus-2 (HSV-2) and human papillomavirus (HPV).

DETAILED DESCRIPTION:
STUDY DESCRIPTION:

The study is being carried out by the Rakai Health Sciences Program, a research collaboration between the Uganda Virus Research Institute/Uganda Ministry of Health, Johns Hopkins Bloomberg School of Public Health and researchers from Makerere University, Kampala, Uganda.

* The study, being conducted in Rakai District, Uganda, has enrolled 997 HIV+ and following a detailed informed consent process, randomizing them to receive either immediate (within several days or weeks) or delayed (two years) circumcision. The goals are to assess the safety and acceptability of male circumcision among HIV+ men, and to assess potential effects of male circumcision on the acquisition of STDs such as HSV-2. Hypotheses are that male circumcision will be acceptable to and safe in HIV+ men, will reduce the rate of acquisition of STDs, and will reduce the frequency of STD symptoms, such as genital ulceration.
* The study has also enrolled 500 men who, regardless of their HIV status, decline to receive their HIV results, despite encouragement to do so. Hypotheses are that circumcision will be acceptable and safe in men who decline their HIV results, and will reduce the rate of acquisition of HIV and STDs, and the frequency of STD symptoms such as genital ulcers.
* The study has enrolled 3,700 female partners of the men in groups 1 and 2 above, as well as of 5,000 HIV-negative men enrolled in a complementary NIH-funded study of male circumcision for HIV prevention (U1 AI51171 which is being separately registered). Following informed consent, the women partners are being followed annually to assess the acceptability and safety of male circumcision in female partners, and potential effects of male circumcision on HIV and STD acquisition. The hypotheses are that male circumcision will be acceptable to and safe in women partners, and will reduce the acquisition of HIV and STDs such as HSV-2 and HPV (human papilloma virus which causes cervical cancer.)
* Finally, the study is also following ~3,000 men and women in the ~50 communities where the circumcision trials are taking place, in order to assess community attitudes towards and knowledge of male circumcision, and to assess whether other preventive behaviors (abstinence, monogamy, numbers of partners, condom use, etc...) change in the community once circumcision becomes available. The hypothesis is that male circumcision will be acceptable in the community and will not result in behavioral disinhibition (increased rates of high risk behaviors).

The Gates-funded study being registered here is complementary to a separate NIH-funded trial of male circumcision in HIV-negative men who accept their HIV results, being carried out by the Rakai Health Sciences Program study team. The latter study, which is enrolling 5000 HIV-negative men, is designed to answer whether male circumcision is acceptable and safe in HIV-neg men, and whether the procedure reduces the acquisition of HIV and STDs.

The complementary Gates-funded trial is designed to answer the following additional questions:

* Is male circumcision acceptable to and safe in HIV-infected men, and will it reduce the rates of acquisition of STDs in these men?

These questions are of great importance for future circumcision programs:

* Will such programs need to screen out HIV+ men (if circumcision is shown to be unsafe in such men, potentially as a result of delayed healing) or should future programs include HIV+ men, if the procedure is safe in them, and has potential benefits such as reduced STD acquisition, improved genital hygiene and reduced rates of STD symptomatology?
* Is male circumcision acceptable and safe in men who decline their HIV results, and will it reduce rates of acquisition of HIV and STDS in these men?

From prior Rakai Program data, the researchers know that men who decline their HIV results tend to have higher risk behaviors. Determining potential circumcision risks in these men (such as, potentially delayed healing because of their higher risk behaviors) or benefits (such as potentially, reduced rates of HIV and STD acquisition) is thus very important for the design of any future large scale circumcision programs. From the public health viewpoint, it will be important to know whether such programs should include or exclude men who decline HIV results. (Please note: the Rakai Program strongly recommends and encourages the receipt of HIV results, and provides the results confidentially and free of charge. The great majority of Rakai Program research participants (85-90%) accept their HIV results, but a minority continue to decline, although the latter group is getting smaller every year. In addition, please also note that even if participants decline their HIV results, the Rakai Program still provides them with detailed HIV prevention education and counseling.) Enrollment of men who decline their HIV results is also congruent with Ugandan Ministry of Health Policy, which encourages but does not force individuals and study participants to receive their HIV results.

Enrollment of female partners is designed to answer important questions regarding potential effects of male circumcision on women. Should male circumcision reduce HIV and STD acquisition in women, this would represent an additional important public health benefit of the procedure and would add to the cost effectiveness of male circumcision programs. However, if the procedure is associated with increased HIV transmission (for example, due to increased transmission before a circumcision surgical would is fully healed), it is crucial that such a potential risk be identified rapidly within a trial, in order to prevent the risk within trials and in any potential future circumcision programs.

Following enrollment, men in the circumcision arm are followed post-operatively at weekly intervals until wound healing is fully certified, , at 4-6 weeks, 6 months, 12 months and 24 months. Men in the control arm are followed at 4-6 weeks and 6, 12 and 24 months. At baseline and follow up, men respond to a detailed sociodemographic, behavioral and health questionnaire, and provide biological samples (venous blood, urine, sub-preputial swabs [prior to circumcision] and for circumcised men, foreskins are collected at time of surgery.) Samples will allow assessment of multiple infections, including HIV, HSV-2, gonorrhea, chlamydia and syphilis.

Women partners are followed annually, through the Rakai Community Cohort Study. Following written informed consent, women are administered a detailed sociodemographic, behavioral and health status questionnaire, and provide venous blood and self-administered vaginal swabs at baseline and study follow up visits. The samples will allow assessment of multiple infections and conditions, including HIV, syphilis, gonorrhea, chlamydia, trichomonas, bacterial vaginosis, HSV-2 and HPV. Women partners of HIV+ men receive additional visita at 6 and 18 months post enrollment.

Community members (men not in the trials, and women who are not partners of men in the trials) are followed annually through the Rakai Community Cohort Study.

Services offered by the Rakai Program to all study participants include HIV and STD prevention education (information on behavioral risk factors and on abstinence, monogamy, being faithful and condom use), free condoms, free HIV counseling and testing for individuals and couples, free STD treatment, access to Rakai Program clinics for general health care, access to Rakai clinics for free HIV antiretroviral (ARV) drug screening and services, prophylaxis for opportunistic infections and nevirapine services for the prevention of mother-to-child HIV transmission. Please note: residents in the 50 villages where the circumcision trials are being conducted have access to Rakai clinics and ARV services whether or not they consent to be in Rakai studies, in order to avoid undue pressure to participate.

ELIGIBILITY:
Inclusion Criteria:

MALES randomized to circumcision:

* Age 15-49
* Able and willing to provide written informed consent
* Have no medical contraindications to male circumcision

FEMALE partners:

* Able and willing to provide written informed consent
* No age limit

Exclusion Criteria:

* Medical contraindications, including penile pathology or anemia (males). Unable or unwilling to provide informed consent.

Please note: for participants under age 18, the study follows informed consent/assent procedures as required under US Federal Regulations. The latter are also consistent with Ugandan policy.

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5200 (Actual)
Dates: Start 2003-08; Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Rates of HIV acquisition in HIV-negative (neg) males and HIV-neg female partners
Rates of STD acquisition in HIV-neg and HIV positive (+) males and HIV-neg and HIV+ female partners

SECONDARY OUTCOMES:
Circumcision safety in HIV+ and HIV-neg males
Behaviors among males and females in couples where the male is randomized to immediate versus delayed circumcision
Behaviors among men and women in the general community

CONTACTS AND LOCATIONS:
Overall Officials: David Serwadda, MBChB,MPH, Principal Investigator — Makerere University Institute of Public Health, Kampala; Godfrey Kigozi, MBChB, MPH, Study Director — Rakai Health Sciences Program
Locations (1):
- Rakai Health Sciences Program, Kalisizo, Rakai District, Uganda

REFERENCES:
- [Derived] Tobian AA, Kong X, Wawer MJ, Kigozi G, Gravitt PE, Serwadda D, Eaton KP, Nalugoda F, Quinn TC, Gray RH. Circumcision of HIV-infected men and transmission of human papillomavirus to female partners: analyses of data from a randomised trial in Rakai, Uganda. Lancet Infect Dis. 2011 Aug;11(8):604-12. doi: 10.1016/S1473-3099(11)70038-X. Epub 2011 Apr 12. PMID 21489882
- [Derived] Wawer MJ, Tobian AA, Kigozi G, Kong X, Gravitt PE, Serwadda D, Nalugoda F, Makumbi F, Ssempiija V, Sewankambo N, Watya S, Eaton KP, Oliver AE, Chen MZ, Reynolds SJ, Quinn TC, Gray RH. Effect of circumcision of HIV-negative men on transmission of human papillomavirus to HIV-negative women: a randomised trial in Rakai, Uganda. Lancet. 2011 Jan 15;377(9761):209-18. doi: 10.1016/S0140-6736(10)61967-8. Epub 2011 Jan 6. PMID 21216000
- [Derived] Serwadda D, Wawer MJ, Makumbi F, Kong X, Kigozi G, Gravitt P, Watya S, Nalugoda F, Ssempijja V, Tobian AA, Kiwanuka N, Moulton LH, Sewankambo NK, Reynolds SJ, Quinn TC, Oliver AE, Iga B, Laeyendecker O, Gray RH. Circumcision of HIV-infected men: effects on high-risk human papillomavirus infections in a randomized trial in Rakai, Uganda. J Infect Dis. 2010 May 15;201(10):1463-9. doi: 10.1086/652185. PMID 20370481
- [Derived] Gray RH, Serwadda D, Tobian AA, Chen MZ, Makumbi F, Suntoke T, Kigozi G, Nalugoda F, Iga B, Quinn TC, Moulton LH, Laeyendecker O, Reynolds SJ, Kong X, Wawer MJ. Effects of genital ulcer disease and herpes simplex virus type 2 on the efficacy of male circumcision for HIV prevention: Analyses from the Rakai trials. PLoS Med. 2009 Nov;6(11):e1000187. doi: 10.1371/journal.pmed.1000187. Epub 2009 Nov 24. PMID 19936044
- [Derived] Wawer MJ, Makumbi F, Kigozi G, Serwadda D, Watya S, Nalugoda F, Buwembo D, Ssempijja V, Kiwanuka N, Moulton LH, Sewankambo NK, Reynolds SJ, Quinn TC, Opendi P, Iga B, Ridzon R, Laeyendecker O, Gray RH. Circumcision in HIV-infected men and its effect on HIV transmission to female partners in Rakai, Uganda: a randomised controlled trial. Lancet. 2009 Jul 18;374(9685):229-37. doi: 10.1016/S0140-6736(09)60998-3. PMID 19616720
- [Derived] Kiggundu V, Watya S, Kigozi G, Serwadda D, Nalugoda F, Buwembo D, Settuba A, Anyokorit M, Nkale J, Kighoma N, Ssempijja V, Wawer M, Gray RH. The number of procedures required to achieve optimal competency with male circumcision: findings from a randomized trial in Rakai, Uganda. BJU Int. 2009 Aug;104(4):529-32. doi: 10.1111/j.1464-410X.2009.08420.x. Epub 2009 Apr 21. PMID 19389002
- [Derived] Tobian AA, Serwadda D, Quinn TC, Kigozi G, Gravitt PE, Laeyendecker O, Charvat B, Ssempijja V, Riedesel M, Oliver AE, Nowak RG, Moulton LH, Chen MZ, Reynolds SJ, Wawer MJ, Gray RH. Male circumcision for the prevention of HSV-2 and HPV infections and syphilis. N Engl J Med. 2009 Mar 26;360(13):1298-309. doi: 10.1056/NEJMoa0802556. PMID 19321868
- [Derived] Tobian AA, Charvat B, Ssempijja V, Kigozi G, Serwadda D, Makumbi F, Iga B, Laeyendecker O, Riedesel M, Oliver A, Chen MZ, Reynolds SJ, Wawer MJ, Gray RH, Quinn TC. Factors associated with the prevalence and incidence of herpes simplex virus type 2 infection among men in Rakai, Uganda. J Infect Dis. 2009 Apr 1;199(7):945-9. doi: 10.1086/597074. PMID 19220138
- [Derived] Kigozi G, Gray RH, Wawer MJ, Serwadda D, Makumbi F, Watya S, Nalugoda F, Kiwanuka N, Moulton LH, Chen MZ, Sewankambo NK, Wabwire-Mangen F, Bacon MC, Ridzon R, Opendi P, Sempijja V, Settuba A, Buwembo D, Kiggundu V, Anyokorit M, Nkale J, Kighoma N, Charvat B. The safety of adult male circumcision in HIV-infected and uninfected men in Rakai, Uganda. PLoS Med. 2008 Jun 3;5(6):e116. doi: 10.1371/journal.pmed.0050116. PMID 18532873